CLINICAL TRIAL: NCT04869787
Title: A Multi-Center, Pilot Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device (SCD) for the Treatment of Immunomodulatory Dysregulation Due to Pediatric Acute Kidney Injury (AKI)
Brief Title: A Multi-Center Study of a SCD for Immunomodulatory Dysregulation in Pediatric AKI
Acronym: SCD PED-02
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The device manufacturer has received a HDE for this population from the FDA
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Stuart Goldstein, MD, Director, Center for Acute Care Nephrology, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCD PED-02
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SCD Treatment (Other): Pediatric patients receiving SCD + CRRT for up to 10 days
  Interventions: Device: Selective Cytopheretic Device

INTERVENTIONS:
Device: Selective Cytopheretic Device — SCD in line with CRRT extracorporeal device
  Other Names: SCD-F40

SUMMARY:
The SCD PED-02 trial is examining the safety and efficacy of the Selective Cytopheretic Device (SCD) in treating pediatric acute kidney injury (AKI). AKI promotes a systemic inflammatory response syndrome (SIRS) which results in systemic microvascular damage and, if severe, multi-organ dysfunction. Activated circulating leukocytes play a central role in this process. The SCD is a synthetic membrane with the ability to bind activated leukocytes and, when used in a continuous renal replacement therapy (CRRT) extracorporeal circuit in the presence of regional citrate anticoagulation, modulates inflammation. The SCD PED-02 study will test the primary hypothesis that up to ten sequential 24-hour SCD treatments in pediatric patients with AKI will be completed safely and improve survival compared to historical controls who received CRRT alone.

DETAILED DESCRIPTION:
The SCD PED-02 trial is examining the safety and efficacy of the Selective Cytopheretic Device (SCD) in treating pediatric acute kidney injury (AKI). Importantly, acute kidney injury is a highly lethal condition in critically ill patients. Despite improvements in acute medical care and advances in dialysis therapies, the mortality rate during the past four decades of this condition has not improved. Critically ill patients with AKI in hospital ICU settings have mortality rates of approximately 50%, including pediatric patients. AKI promotes a systemic inflammatory response syndrome (SIRS) which results in systemic microvascular damage and, if severe, multi-organ dysfunction. Activated circulating leukocytes play a central role in this process. Leukocytes, especially neutrophils, are major contributors to the pathogenesis and progression of many inflammatory disorders, including SIRS, sepsis, ischemia reperfusion injury, and acute respiratory distress syndrome (ARDS). Many therapeutic approaches are under investigation to limit the activation and tissue accumulation of leukocytes at sites of inflammation to minimize tissue destruction and disease progression.

The SCD is comprised of tubing, connectors, and a synthetic membrane cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and it is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits. The SCD is a synthetic membrane with the ability to bind activated leukocytes and, when used in a continuous renal replacement therapy (CRRT) extracorporeal circuit in the presence of regional citrate anticoagulation, modulates inflammation.

The SCD PED-02 study will test the primary hypothesis that up to ten sequential 24-hour SCD treatments in pediatric patients with AKI will be completed safely and improve survival compared to historical controls who received CRRT alone.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's parent or legal representative has provided informed consent
2. Must be receiving medical care in an intensive care unit
3. Age less than 18 years.
4. Body weight between ≥10 and ≤ 20 kilograms
5. Intent to receive full supportive care through aggressive management
6. Clinical diagnosis of AKI requiring CRRT
7. At least one non-renal organ failure OR presence of proven/suspected sepsis

Exclusion Criteria:

1. Threshold blood pressure of 80/40 mmHg
2. Patients with a solid organ transplant or those with a bone marrow or stem cell transplant in the previous 100 days or who have not engrafted
3. Acute or chronic use of circulatory support device, other than extracorporeal membrane oxygenation (ECMO)
4. Presence of preexisting advanced chronic renal failure on chronic renal replacement therapy or with an estimated glomerular filtration rate less than 30 mL/min/1.73m2
5. AKI occurring in the setting of burns, obstructive uropathy, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, cyclosporine or tacrolimus nephrotoxicity
6. Metastatic malignancy which is actively being treated or may be treated by chemotherapy or radiation during the subsequent three month period after study therapy
7. Chronic immunosuppression with the exception of corticosteroids up to a dose of 10 mg of prednisone per day
8. Known positive HIV or AIDS or COVID-19
9. Current Do not Attempt Resuscitation (DNAR), Allow Natural Death (AND), or withdrawal of care status, or anticipated change in status within the next 7 days
10. Patient not expected to survive 28 days because of an irreversible medical condition
11. Any medical condition that the Investigator thinks may interfere with the study objectives
12. Treating clinician does not feel it is in the best interest of the patient
13. Platelet count <15,000/mm3
14. Concurrent enrollment in another interventional clinical trial
15. Use of any other investigational drug or device within the previous 30 days
16. Use of AN-69 hemofilter membrane for CRRT

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's of Alabama, Birmingham, Alabama
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After consent was obtained, participants entered the screening period. If their clinical status changed and the investigator believed that they no longer met eligibility criteria, the participant would be recorded as a screen failure. Criteria this may impact included resuscitation status, hypotension, platelet count, medical condition that the investigator thought would interfere with study objectives. or treating physician believed it was not longer in the patient's best interest.
Period: Screening
Arm/Group | SCD Treatment
Started | 7
Completed | 6
Not Completed | 1
Not completed — Physician Decision | 1
Period: SCD Treatment Period (up to 10 Days)
Arm/Group | SCD Treatment
Started | 6
Completed | 5
Not Completed | 1
Not completed — Death | 1
Period: Observational Follow Up Period (90 Days)
Arm/Group | SCD Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who went on to receive treatment with the SCD
Arm/Group | SCD Treatment
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.05 [1.77 to 3.48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Body Weight, Continuous [Median (Inter-Quartile Range); unit: kilograms] | 13.4 [12.0 to 14.1]
Pediatric Risk of Mortality II Score [Median (Inter-Quartile Range); unit: Scores on a scale] — The PRISM II (Pediatric Risk of Mortality) score was created and published by Dr. M. Pollack in 1988 as a way to objectively measure severity of illness of critically ill pediatric patients. In this research study, the PRISM II was calculated in the 12 hours immediately prior to the initiation of the investigational device therapy. The algorithm measures 14 physiologic variables to create the PRISM score with a range from 0 to 76, with a higher score equating to a higher risk of death.
  Scores on a scale | 16.5 [14 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Number of SCD-related Adverse Events (AE)
Description: Total number of AEs across all participants that are considered to be at least possibly related to SCD therapy per the site investigator
Time Frame: From enrollment to Day 60 post treatment
Population: Participants who received treatment with the SCD
Measure: Number; unit: Events
Arm/Group | SCD Treatment
Number analyzed (Participants) | 6
Events | 1

2. Primary Outcome: Number of Unanticipated Adverse Device Effects (UADE)
Description: Total number of UADEs across all participants treated with the SCD
Time Frame: From enrollment to Day 60 post treatment
Population: Participants who received treatment with the SCD
Measure: Number; unit: Events
Arm/Group | SCD Treatment
Number analyzed (Participants) | 6
Events | 0

3. Secondary Outcome: Mortality
Description: Mortality rate as a percent of all participants treated with the SCD
Time Frame: Day 28 post treatment
Population: Participants who received treatment with the SCD
Measure: Count of Participants; unit: Participants
Arm/Group | SCD Treatment
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Renal Recovery
Description: Percent of patients free from chronic dialysis treatments
Time Frame: Day 28 post treatment
Population: Participants who received treatment with the SCD and who survived to Day 28 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | SCD Treatment
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Hospital Length of Stay
Description: Total days each participant spends as an inpatient at an acute care facility
Time Frame: From enrollment to Day 60 post treatment
Population: Participants who received treatment with SCD, survived to hospital discharge, and were discharged prior to the last study visit (Day 60)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | SCD Treatment
Number analyzed (Participants) | 2
Days | 24 [23 to 25]

6. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: Total days each participant spends in an ICU during the primary admission
Time Frame: From enrollment to Day 60 post treatment
Population: Participants who received treatment with the SCD, survived to Day 60, and were ICU discharged by the last study visit (Day 60)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | SCD Treatment
Number analyzed (Participants) | 4
Days | 11.5 [10 to 24]

7. Secondary Outcome: Mortality
Description: Mortality rate as a percent of all participants treated with the SCD
Time Frame: Day 60 post treatment
Population: Participants who received treatment with the SCD
Measure: Count of Participants; unit: Participants
Arm/Group | SCD Treatment
Number analyzed (Participants) | 6
Participants | 1

8. Secondary Outcome: Renal Recovery
Description: Percent of patients free from chronic dialysis treatments
Time Frame: Day 60 post treatment
Population: Participants who received treatment with the SCD and who survived to Day 60 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | SCD Treatment
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 60 Days
Description: During the screening period, only adverse events directly related to screening procedures were captured. Serious adverse events were monitored for and collected between SCD start and Day 60 after enrollment for each participants. Non-serious adverse events were recorded from SCD start until 120 hours after SCD treatment ends, death, subject withdrawal of study consent, or ICU discharge, whichever occurs first.
Arm/Group | SCD Treatment
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCD Treatment (N=6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Medical device site thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCD Treatment (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Cerebral dysfunction (Nervous system disorders) | 1 (1)
Device leakage (Product Issues) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was terminated early in preparations for a HDE approval from the FDA for this population. This trial represents a small subject populations from only 2 centers in the US.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT04869787/Prot_SAP_000.pdf